CLINICAL TRIAL: NCT04555824
Title: A Randomized, Double-blind, Placebo-Controlled, Single Dose,Dose-escalation，Phase 1a Study of the Safety, Tolerability，Pharmacokinetics and the Potential Immunological Reaction of Recombinant Human Thymosin Beta4 in Chinese Healthy Volunteers
Brief Title: A Phase 1a Study of Thymosin Beta 4 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL005-Ⅰ-2015-1
Record Dates: First submitted 2018-09-14; First posted 2020-09-21 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Recombinant human thymosin β4

STUDY DESIGN:
Intervention Model Description: Dose Escalation for 7 Cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Recombinant Human Thymosin β4 Dose 1 group (Experimental): Two subjects in this group will receive NL005 for 0.05ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Dose 2 groupRecombinant Human Thymosin β4 (Experimental): Two subjects in this group will receive NL005 for 0.25ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Dose 3 groupRecombinant Human Thymosin β4 (Experimental): Eight subjects in this group will receive NL005 for 0.5ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Dose 4 groupRecombinant Human Thymosin β4 (Experimental): Eight subjects in this group will receive NL005 for 2ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Dose 5 groupRecombinant Human Thymosin β4 (Experimental): Eight subjects in this group will receive NL005 for 5ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Recombinant Human Thymosin β4 Dose 6 group (Experimental): Eight subjects in this group will receive NL005 for 12.5ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Recombinant Human Thymosin β4 Dose 7 group (Experimental): Eight subjects in this group will receive NL005 for 25ug/kg respective in D1.
  Interventions: Drug: Recombinant Human Thymosin β4
- Placebo (Placebo Comparator): Two subjects in each dose group（0.5/2/5/12.5/25ug/kg）were given placebo respective in D1. A total of 10 subjects were given placebos.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Recombinant Human Thymosin β4 — Healthy subjects , were given a single intravenous dose of rh-Tβ4 in Day1.
  Other Names: rh-β4
  Arms: Dose 2 groupRecombinant Human Thymosin β4; Dose 3 groupRecombinant Human Thymosin β4; Dose 4 groupRecombinant Human Thymosin β4; Dose 5 groupRecombinant Human Thymosin β4; Recombinant Human Thymosin β4 Dose 1 group; Recombinant Human Thymosin β4 Dose 6 group; Recombinant Human Thymosin β4 Dose 7 group
Other: Placebo — Five cohorts, with 10 healthy subjects , were given a single intravenous dose of Placebo. Cohorts received ascending doses of either 0.5, 2,5,12.5 or 25 ug/kg in Day1.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerance, pharmacokinetics and the potential immunological reaction of single intravenous recombinant human thymosin β4（NL005）or placebo 0.05, 0.25, 0.5, 2, 5, 12.5, 25μg/kg in Chinese healthy volunteers. 54 volunteers will be randomized to receive NL005 or placebo for 7 cohorts,administered iv by iv push on Day 1.

DETAILED DESCRIPTION:
This study is a randomized,double-blind,placebo-controlled, investigation to evaluate the safety, tolerability, pharmacokinetics and the potential immunological reaction of single of NL005 administered intravenously to healthy volunteers.

In Phase 1A, Seven (7) cohorts of subjects (first two cohorts 2 subjects respectively, 10 subjects per cohort for next 5 cohorts) will administered one dose of NL005 or placebo in a 4:1 ratio. Dosing start at 0.05μg/kg and advance to 0.25, 0.5, 2, 5, 12.5, 25μg/kg.

NL005 or placebo administered as a single dose on Day 1. Safety parameters recorded on Study Days 1, 2, 5, 14, and 28. Evaluation of adverse events performed throughout the study. Pharmacokinetic samples obtained on Study Day 1. Blood samples collected for serum antibody determinations at Screening , Days 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy volunteers（male or female）.
2. Between 18 and 50 years of age.
3. BMI between 19 and 28 kg/m2.
4. Good health condition, no history of unintentional, liver, kidney, digestive tract, immune system, nervous system, mental and metabolic abnormality, no family history of tumor.
5. Medical history , physical examination, laboratory examinations are normal or not clinically significant abnormalities, and the investigator judges those who are qualified.
6. Voluntarily sign informed consent.

Exclusion Criteria:

1. Physical examination, vital signs, ECG or laboratory examinations are abnormal (clinically significant ).
2. Active hepatitis b or c patients, carriers of hepatitis b virus.
3. HIV antibody test positive or syphilis spiral antibody test positive.
4. ADA tests positive.
5. Smoke more than 5 cigarettes a day, had a suspected or proven history of substance abuse, and consumed an average of more than 2 units of alcohol per day for 3 months (1 unit =12 ounces or 360mL beer, 5 ounces or 150mL liquor, 1.5 ounces or 45mL distilled liquor) or had a positive alcohol test.
6. Participated in another trial or used this drug within 3 months before inclusion.
7. Any other drug was used within two weeks before the trial.
8. There is a significant clinical history of allergy, especially for drugs, protein preparations and biological products, especially for rh-tβ4 or any of its ingredients.
9. Blood donation or blood loss was equal to or greater than 400 mL within three months prior to the trial.
10. Women who are pregnant or breast-feeding, or who are likely to become pregnant and do not use an acceptable method of contraception, or who have a positive pregnancy test and who do not use effective contraception or whose partner plans to give birth within six months.
11. Unable to tolerate venous blood collection.
12. There is no guarantee that smoking and taking grapefruit juice or any alcoholic and xanthine food and beverage (including chocolate, tea, coffee, cola, etc.) from 48 hours before administration to the last blood sample collection.
13. The investigator judges that the subject is unable to complete the study or otherwise considers that the subject's participation in the study may cause other injury.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) . | Day1
  Determine maximum tolerated dose (MTD) or dose-limiting toxicity (DLT) by comprehensive evaluation of drug safety by adverse event observation, vital signs, physical examination, laboratory examination, electrocardiogram, etc. In this study, DLT was defined as liver, kidney, heart and mental nervous system toxicity of level 2 or above or blood system toxicity of level 3 or above and other systemic adverse events occurred within 14 days after drug administration, and the adverse events were judged to be related to the experimental drug use.If more than 3 (including 3) DLT cases are present in any dose group, the test should be terminated. The previous dose of this dose is considered the maximum tolerated dose (MTD).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | Day1
  Determine maximum tolerated dose (MTD) or dose-limiting toxicity (DLT) by comprehensive evaluation of drug safety by adverse event observation, vital signs, physical examination, laboratory examination, electrocardiogram, etc. All adverse events were determined according to NCI CTCAE4.03.CTCAE4.03 was classified into grades 1 to 5, in which grade 1 was mild adverse event and grade 5 was death due to adverse event.
The Cmax of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The Tmax of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The MRT of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The AUClast of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The AUC0-inf of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The t1/2 of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The VZ of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The CL of single ascending doses of rh-Tβ4. | Day 1.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , Tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The potential immunological reaction (antibody formation) of single ascending doses of rh-Tβ4. | Day 1、14、28.
  Approximately 5mL venous blood was collected from subjects before, 14 days after, and 28 days after administration for ADA study of rh-Tβ4 in healthy subjects.After the 28th-day follow-up period, subjects who confirm that ADA results are positive should be reexamined every 30 days (±3 days) until the results turn negative or the titer level is stable for two consecutive times.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Beijing, China

REFERENCES:
- See also: Related Info — http://www.northland-bio.com/